CLINICAL TRIAL: NCT01572935
Title: Body Weight Assessment in Swiss Primary School Children: Trend Analysis Over 10 Years
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr. med., Swiss Federal Institute of Technology
Other Study IDs: EK 2011-N-50
Record Dates: First submitted 2012-02-08; First posted 2012-04-06 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Overweight; Obesity
Keywords: childhood obesity prevalence
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Recent evidence from several countries has emerged suggesting that the increase in the prevalence of childhood obesity has slowed down substantially, or even leveled off. Also in Switzerland this trend has been observed. In 2002, 20.3% and 19.1% of boys and girls, respectively, were overweight or obese in Switzerland. In 2007, the prevalence of overweight was significantly lower, with 11.3% and 9.9% of school-aged boys and girls, respectively, being overweight or obese. Further trend analyses are necessary to confirm that the stabilizing trend observed reflects a long-term change in the rates of childhood overweight and obesity.

Objective and Methods: The aim of the present study is to repeat the 2002 and 2007 national studies, in order to monitor the trend in the prevalence of overweight and obesity in 6-12 year old children in Switzerland during this 5 respectively 10 year time period. Height and weight will be measured and used to calculate body mass index (BMI). BMI references form the Centers for Disease Control and Prevention will be used to determine the prevalence of underweight (< 5th percentile), overweight (≥ 85th and < 95th percentile) and obesity (≥ 95th percentile). Waist and hip circumference will be measured. Moreover, skinfold thicknesses and bioelectrical impedance analysis will be performed to calculate body fat percentage.

ELIGIBILITY:
Inclusion Criteria:

* age 6-12 years
* child is attending one of the selected classrooms

Exclusion Criteria:

* age below 6 or above 12 years

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 3 classrooms each from 60 randomly selected schools
Sampling Method: Probability Sample
Enrollment: 2979 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of overweight and obesity | up to 7 months
  Assessment of the prevalence of overweight and obesity in the study population using measurements of weight and height to calculate the body mass index. The 85th and 95th percentiles of the reference population published by the Centers for Disease Control and Prevention will be used as cut-off points.

SECONDARY OUTCOMES:
Waist circumference | up to 7 months
  Assessment of waist circumference using non-strechable measuring tape.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Prof, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Aeberli I, Henschen I, Molinari L, Zimmermann MB. Stabilization of the prevalence of childhood obesity in Switzerland. Swiss Med Wkly. 2010 Jul 15;140:w13046. doi: 10.4414/smw.2010.13046. eCollection 2010. PMID 20349364
- [Background] Zimmermann MB, Gubeli C, Puntener C, Molinari L. Overweight and obesity in 6-12 year old children in Switzerland. Swiss Med Wkly. 2004 Sep 4;134(35-36):523-8. doi: 10.4414/smw.2004.10640. PMID 15517505
- [Background] Aeberli I, Ammann RS, Knabenhans M, Molinari L, Zimmermann MB. Decrease in the prevalence of paediatric adiposity in Switzerland from 2002 to 2007. Public Health Nutr. 2010 Jun;13(6):806-11. doi: 10.1017/S1368980009991558. Epub 2009 Sep 22. PMID 19772692